CLINICAL TRIAL: NCT01205191
Title: Effectiveness Study of Cell Phone-supported Cognitive Behavioural Therapy for Anxiety Disorders in Frontline Settings
Brief Title: Cell Phone-supported Cognitive Behavioural Therapy
Acronym: LINNEA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Toomas Timpka, professor, Section of Social Medicince/LiU
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LFP5/08
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-09

CONDITIONS: Anxiety
Keywords: Cognitive behavioural therapy; Anxiety; Primary care; Effectiveness trial; Cell-phone supported therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBT-ubiquitous (Experimental)
  Interventions: Behavioral: Cell-phone supported CBT
- CBT-placebo (Placebo Comparator): Cognitive behavioural therapy provided with access to a digital audio player with self-administered materials for stress management
  Interventions: Behavioral: CBT with digital audio player support
- CBT-TAU (Active Comparator): Cognitive behavioural Therapy provided 'As Usual'
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: Cell-phone supported CBT — Cognitive behavioural therapy provided with all-time (ubiquitous) support by cell phone applications
  Arms: CBT-ubiquitous
Behavioral: CBT with digital audio player support — Cognitive behavioural therapy provided with access to a digital audio player with self-administered materials for stress management and relaxation.
  Arms: CBT-placebo
Behavioral: CBT — CBT for anxiety disorders
  Arms: CBT-TAU

SUMMARY:
Definitions

CBT-ubiquitous - Cognitive behavioural therapy (CBT) provided with all-time (ubiquitous) support by cell phone applications CBT-TAU - Cognitive behavioural Therapy provided 'As Usual' CBT-placebo - Cognitive behavioural therapy provided with access to a digital audio player with self-administered materials for stress management and relaxation.

Study objectives

1. to compare the relative effectiveness of a computerized ubiquitous CBT (CBT-ubiquitous) against anxiety disorders with CBT-treatment as usual (CBT-TAU);
2. to assess the safety and tolerability of the CBT-ubiquitous as compared with CBT-TAU and CBT provided with access to a placebo technical device (CBT-placebo)..

Study implementation

The investigators hypothesize that all active treatments are superior to placebo given evidence that face-to-face CBT is effective in the treatment of both anxiety and depression. The investigators also predict that patients receiving CBT-ubiquitous will show greater improvement than those given CBT-TAU, and assume that CBT-ubiquitous leads to improved adherence with treatment compared to CBT-TAU and CBT-placebo.

The investigators will use an intention to treat (ITT) approach to fulfill the study aims, by which the investigators mean that clients are analysed as randomized rather than by treatment actually received. The study will be implemented in the central district of Östergötland County Council (pop 145.000). The research group has in two previous projects (VINNOVA 2005-2007, VINNOVA 2008-2009) established cooperation with the 'Unga Vuxna' (Young Adults) service provided in this district. The service supplies CBT to the subpopulation experiencing early stages of mental disorders in the age group 16-25 years (n=20,000) in order to prevent development of significant psychiatric disease and disability. The service employs six therapists with at least one year specific CBT training and is co-located with Primary Healthcare Centres (PHCs) in downtown Linköping, Åtvidaberg and Kisa. Clients staying outside the urban areas can make appointments with therapists at their closest PHC on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 25; and
* scoring 7 or higher on the anxiety section of the Hospital Anxiety and Depression scale (HADS) at initial evaluation.

Exclusion Criteria:

* at the initial evaluation displays symptoms indicative for referral to a psychiatric specialist, e.g. active suicidal ideas or symptoms of a psychotic disorder, organic mental disorder or alcohol and/or drug dependence; or
* is unable to read, write or speak in the Swedish;

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Six months after treatment
  Hospital Anxiety and Depression Scale-Anxiety (HADS-A), General Health Questionnaire-12 (GHQ-12), Beck's Anxiety Index (BAI)

SECONDARY OUTCOMES:
Adherence | 14 weeks
  Data is collected from the therapists on whether the client has
  * discontinued the CBT program by not showing up at sessions;
  * discontinued the CBT program by actively informing the therapist;
  * been discontinued from the treatment by the therapist;
  * fulfilled the "therapeutic contract", e.g. by completing 'homework' agreed upon.

CONTACTS AND LOCATIONS:
Overall Officials: Toomas Timpka, MD PhD, Principal Investigator — Section of Social Medicine/LiU
Locations (1):
- "Unga Vuxna" Clinic, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Ekberg J, Timpka T, Bang M, Froberg A, Halje K, Eriksson H. Cell phone-supported cognitive behavioural therapy for anxiety disorders: a protocol for effectiveness studies in frontline settings. BMC Med Res Methodol. 2011 Jan 10;11:3. doi: 10.1186/1471-2288-11-3. PMID 21219593